CLINICAL TRIAL: NCT04944784
Title: A Phase 3, Multi-Center, Double-Blind, Randomized, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Reldesemtiv in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Study to Evaluate the Efficacy and Safety of Reldesemtiv in Patients With Amyotrophic Lateral Sclerosis (ALS)
Acronym: COURAGE-ALS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The DMC recommended the trial be discontinued due to futility following a planned second interim analysis.
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CY 5031; 2020-004040-29 (EudraCT Number)
Record Dates: First submitted 2021-06-16; First posted 2021-06-30 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; CK-2127107; Reldesemtiv; COURAGE-ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — reldesemtiv

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Reldesemtiv Group, Double-Blind Period (Experimental): Participants in this arm take 2 reldesemtiv 150 mg oral tablets twice a day for a 600 mg total daily dose from Day 1 until Week 24.
  Interventions: Drug: Reldesemtiv
- Placebo Group, Double-Blind Period (Placebo Comparator): Participants in this arm take 2 placebo oral tablets twice a day from Day 1 until Week 24.
  Interventions: Drug: Placebo
- Delayed Start Group, Active Drug Period (Experimental): Participants in this arm were those who received placebo in the double-blind period and reldesemtiv in the active drug period. Participants take 2 reldesemtiv 150 mg oral tablets twice a day for a 600 mg total daily dose from Week 24 until Week 48. Patients who were down-titrated for any reason during the 24 weeks of blinded dosing take 1 reldesemtiv 150 mg oral tablet twice a day for a 300 mg total daily dose from Week 24 until Week 48.
  Interventions: Drug: Reldesemtiv
- Early Start Group, Active Drug Period (Experimental): Participants in this arm were those who received reldesemtiv in the double-blind and active drug periods. Participants take 2 reldesemtiv 150 mg oral tablets twice a day for a 600 mg total daily dose from Week 24 until Week 48. Patients who were down-titrated for any reason during the 24 weeks of blinded dosing take 1 reldesemtiv 150 mg oral tablet twice a day for a 300 mg total daily dose from Week 24 until Week 48.
  Interventions: Drug: Reldesemtiv

INTERVENTIONS:
Drug: Reldesemtiv — Reldesemtiv Oral Tablet
  Arms: Delayed Start Group, Active Drug Period; Early Start Group, Active Drug Period; Reldesemtiv Group, Double-Blind Period
Drug: Placebo — Placebo Oral Tablet
  Arms: Placebo Group, Double-Blind Period

SUMMARY:
The purpose of this study is to assess the effect of reldesemtiv versus placebo on functional outcomes in ALS.

DETAILED DESCRIPTION:
COURAGE-ALS is a Phase 3, double-blind, randomized, placebo-controlled trial of reldesemtiv in patients aged 18 to 80 with ALS.

The screening and qualification period for the trial will be no more than 21 days in duration. Approximately 555 eligible ALS patients will be randomized (2:1) to receive the following dose of reldesemtiv or placebo (stratified by riluzole use/non-use and edaravone use/non-use) for the first 24 weeks (double-blind, placebo-controlled period):

* 300 mg reldesemtiv twice a day for a 600 mg total daily dose (TDD)
* Placebo twice daily

At the end of the 24-week double-blind, placebo-controlled period, patients will transition to the active drug period, where all patients will receive the following dose of reldesemtiv for the next 24 weeks:

* 300 mg reldesemtiv twice a day for a 600 mg TDD for patients who were not down titrated during the 24 weeks of blinded dosing
* 150 mg reldesemtiv twice a day for a 300 mg TDD for patients who were down titrated during the 24 weeks of blinded dosing

ELIGIBILITY:
Key Inclusion Criteria:

* Males or Females between the ages of 18 and 80 years of age, inclusive
* Diagnosis of familial or sporadic ALS (defined as meeting the laboratory-supported probable, probable, or definite criteria for ALS according to the World Federation of Neurology El Escorial criteria). Patients who meet the possible criteria are eligible if they have lower motor neuron findings; those who have purely upper motor neuron findings are ineligible.
* First symptom of ALS ≤ 24 months prior to screening. The qualifying first symptoms of ALS are limited to manifestations of weakness in extremity, bulbar, or respiratory muscles.
* ALSFRS-R total score ≤ 44 at screening. Patients with a total score of 45 or higher may be rescreened 60±7 days following the original screening date.
* Upright FVC ≥ 65.0% of predicted for age, height, sex and ethnicity at screening according to Global Lung Initiative equation
* Must be either on riluzole for ≥ 30 days prior to screening or have not taken it for at least 30 days prior to screening
* Must have completed at least 2 cycles of edaravone at the time of screening or have not received it for at least 30 days prior to screening
* Able to swallow whole tablets

Exclusion Criteria:

* eGFRCysC < 45.0 mL/min/1.73 m2 at screening
* Urine protein/creatinine ratio > 1 mg/mg (113 mg/mmol) at screening
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3-times the upper limit of normal (ULN)
* Total bilirubin (TBL), direct or indirect bilirubin above the ULN.
* Cognitive impairment, related to ALS or otherwise that impairs the patient's ability to understand and/or comply with study procedures and provide informed consent
* Other medically significant neurological conditions that could interfere with the assessment of ALS symptoms, signs or progression.
* Has a tracheostomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cytokinetics, MD, Study Director — Cytokinetics
Locations (84):
- United States (36):
  - St. Joseph's Hospital & Medical Center - Barrow Neurological Institute, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Irvine - ALS & Neuromuscular Center, Orange, California
  - California Pacific Medical Center - Forbes Norris MDA/ALS Research Center, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Colorado Hospital Anschutz Outpatient Pavilion, Aurora, Colorado
  - GW Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Florida Jacksonville, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of South Florida - Carol and Frank Morsani Center for Advanced Health Care, Tampa, Florida
  - Duchossois Center for Advanced Medicine, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Outpatient Center, Baltimore, Maryland
  - Massachusetts General Hospital - Neurological Clinical Research Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center/Medical School, Worcester, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine - Center for Advance Medicine, St Louis, Missouri
  - Neurology Associates, PC, Lincoln, Nebraska
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Atrium Health Neuroscience Institute - Charlotte, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Providence ALS Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center - Clinical Research Center, Nashville, Tennessee
  - Texas Neurology, P.A., Dallas, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - VCU Neuroscience Orthopaedic and Wellness Center (NOW), Henrico, Virginia
  - Froedtert Hospital, Milwaukee, Wisconsin
- Australia (5):
  - Brain and Mind Centre, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Perron Institute, Nedlands, Western Australia
- UZ Leuven Gasthuisberg, Department of Neurology, Leuven, Belgium
- Canada (11):
  - University of Calgary - Heritage Medical Research Clinic, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - McMaster University Medical Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Research Institute - Civic Campus, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Centre de recherche du CHUM, Montreal, Quebec
  - McGill University, Montreal Neurological Institute & Hospital, Montreal, Quebec
  - CHU de Quebec-Université Laval, Québec, Quebec
  - Saskatoon City Hospital, Saskatoon, Saskatchewan
- Deparment of Neurology Bispebjerg University Hospital, Copenhagen, Denmark
- France (7):
  - CRC SLA de Lyon, Bron
  - CHRU de Lille Hopital Roger Salengro, Lille
  - CHU de Limoges - Hopital Dupuytren, Limoges
  - CHU de la Timone, Marseille
  - CHU de Nice - Hôpital Pasteur 2, Nice
  - Hopital La Pitie Salpetriere, Paris
  - CHRU de Tours, Hopital Bretonneau, Clinical Research Center, Tours
- Germany (6):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Medical School Hannover - Department of Neurology, Hanover
  - Universitatsklinikum Jena, Jena
  - Universitätsklinikum Schleswig Holstein, Lübeck
  - Universitatsklinikum Ulm, Ulm
- RSCI Education and Research Centre, Beaumont Hospital, Beaumont, Dublin, Ireland
- Italy (4):
  - Ospedale San Luca, Milan
  - Centro Clinical Nemo - Fondazione Serena Onlus, Milan
  - Instituti Clinici Scientifici Maugeri, Milan
  - AOU Città della Salute e Scienza (Molinette),, Turin
- UMC Utrecht, Department of Neurology, ALS Center, Utrecht, Netherlands
- City Clinic Research, Warsaw, Poland
- Centro Hospitalar Universitario Lisboa Norte, Department of Neurology, Lisbon, Portugal
- Spain (4):
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Basurto, Bilbao
  - Hospital San Rafael, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Neurologimottagningen Skane University Hospital, Malmo
  - Studieenheten Akademiskt Specialistcentrum, Sabbatsberg Hospital, Stockholm
- Muskelzentrum/ALS Clinic, Sankt Gallen, Switzerland
- United Kingdom (2):
  - The Walton Centre NHS Foundation Trust, Liverpool
  - Maurice Wohl Clinical Neuroscience Institute, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rudnicki SA, Giacomelli E, Herder K, Ingre C, Kupfer S, Malik FI, Meng L, Paganoni S, Schellenberg K, Scirocco E, Simkins T, Wei J, Shefner JM; COURAGE-ALS Study Group. The Use of Durable Medical Equipment in COURAGE-ALS, a Phase 3, Multicentre, Randomized Clinical Trial for ALS. Muscle Nerve. 2026 Jan 19. doi: 10.1002/mus.70150. Online ahead of print. PMID 41553108
- [Derived] Rudnicki SA, Gebrehiwet P, Kupfer S, Malik FI, Meng L, Simkins T, Wei J, Wolff AA, Shefner JM. Participant, site personnel and sponsor perspectives on decentralized trial features in COURAGE-ALS: a randomized clinical trial. Amyotroph Lateral Scler Frontotemporal Degener. 2025 Nov;26(7-8):812-820. doi: 10.1080/21678421.2025.2523941. Epub 2025 Jun 27. PMID 40576049
- [Derived] Shefner JM, Cudkowicz ME, Genge A, Hardiman O, Al-Chalabi A, Andrews JA, Chio A, Corcia P, Couratier P, de Carvalho M, Heiman-Patterson T, Henderson RD, Ingre C, Johnston W, Ludolph A, Maragakis NJ, Miller TM, Mora JS, Petri S, Simmons Z, van den Berg LH, Zinman L, Kupfer S, Malik FI, Meng L, Simkins TJ, Wei J, Wolff AA, Rudnicki SA; COURAGE-ALS Study Group. Reldesemtiv in Amyotrophic Lateral Sclerosis: Results From the COURAGE-ALS Randomized Clinical Trial. JAMA Neurol. 2025 May 1;82(5):477-485. doi: 10.1001/jamaneurol.2025.0241. PMID 40126464
- [Derived] Shefner JM, Al-Chalabi A, Andrews JA, Chio A, De Carvalho M, Cockroft BM, Corcia P, Couratier P, Cudkowicz ME, Genge A, Hardiman O, Heiman-Patterson T, Henderson RD, Ingre C, Jackson CE, Johnston W, Lechtzin N, Ludolph A, Maragakis NJ, Miller TM, Mora Pardina JS, Petri S, Simmons Z, Van Den Berg LH, Zinman L, Kupfer S, Malik FI, Meng L, Simkins TJ, Wei J, Wolff AA, Rudnicki SA. COURAGE-ALS: a randomized, double-blind phase 3 study designed to improve participant experience and increase the probability of success. Amyotroph Lateral Scler Frontotemporal Degener. 2023 Aug;24(5-6):523-534. doi: 10.1080/21678421.2023.2216223. Epub 2023 May 30. PMID 37254449

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants were randomized but never dosed in the study.
Period: Double-blind Period
Arm/Group | Reldesemtiv Group, Double-Blind Period | Placebo Group, Double-Blind Period | Delayed Start Group, Active Drug Period | Early Start Group, Active Drug Period
Started | 325 | 161 | 0 | 0
Completed | 180 | 96 | 0 | 0
Not Completed | 145 | 65 | 0 | 0
Not completed — Study Terminated by Sponsor | 96 | 46 | 0 | 0
Not completed — Adverse Event | 20 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 4 | 0 | 0
Not completed — Death | 7 | 2 | 0 | 0
Not completed — Physician Decision | 2 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Sponsor Request | 2 | 1 | 0 | 0
Not completed — Planned Medical Assistance in Dying | 0 | 3 | 0 | 0
Not completed — Participant Choice | 1 | 1 | 0 | 0
Not completed — Progressive Disease | 2 | 2 | 0 | 0
Period: Active Drug Period
Arm/Group | Reldesemtiv Group, Double-Blind Period | Placebo Group, Double-Blind Period | Delayed Start Group, Active Drug Period | Early Start Group, Active Drug Period
Started | 0 | 0 | 96 | 180
Completed | 0 | 0 | 31 | 62
Not Completed | 0 | 0 | 65 | 118
Not completed — Study Terminated by Sponsor | 0 | 0 | 49 | 92
Not completed — Adverse Event | 0 | 0 | 3 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 7
Not completed — Death | 0 | 0 | 3 | 4
Not completed — Lack of Efficacy | 0 | 0 | 2 | 2
Not completed — Planned Medical Assistance in Dying | 0 | 0 | 0 | 1
Not completed — Participant Choice | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 4 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set, which included all enrolled participants, was used for the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Reldesemtiv Group, Double-Blind Period | Placebo Group, Double-Blind Period | Total
Number analyzed (Participants) | 325 | 161 | 486
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The Full Analysis Set, which was used for efficacy outcome measures, was used for the baseline measure analysis population.
  years
    number analyzed (Participants) | 323 | 159 | 482
    (all) | 59.2 (11.00) | 59.8 (10.79) | 59.4 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 64 | 177
  Male | 212 | 97 | 309
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 12 | 27
  Not Hispanic or Latino | 278 | 132 | 410
  Unknown or Not Reported | 32 | 17 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 308 | 149 | 457
  More than one race | 9 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 97 | 56 | 153
  United Kingdom | 0 | 3 | 3
  Switzerland | 2 | 0 | 2
  Portugal | 12 | 3 | 15
  Spain | 29 | 10 | 39
  Canada | 48 | 24 | 72
  Netherlands | 5 | 7 | 12
  Sweden | 8 | 7 | 15
  Belgium | 6 | 1 | 7
  Ireland | 6 | 2 | 8
  Poland | 9 | 7 | 16
  Denmark | 1 | 0 | 1
  Italy | 21 | 11 | 32
  Australia | 22 | 5 | 27
  France | 24 | 14 | 38
  Germany | 35 | 11 | 46
Forced vital capacity (FVC) percent predicted [Mean (Standard Deviation); unit: percent predicted] — Population: Full Analysis Set was used.
  percent predicted
    number analyzed (Participants) | 323 | 159 | 482
    (all) | 84.5 (14.69) | 85.8 (14.19) | 84.9 (14.53)
ALSFRS-R total score [Mean (Standard Deviation); unit: score on a scale] — Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) total score; rating scale 0 to 48; higher scores indicate better functional Population: Full Analysis Set was used.
  score on a scale
    number analyzed (Participants) | 323 | 159 | 482
    (all) | 37.2 (4.97) | 36.6 (5.44) | 37.0 (5.14)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Full Analysis Set was used.
  kg/m^2
    number analyzed (Participants) | 323 | 159 | 482
    (all) | 26.9 (5.67) | 26.4 (4.41) | 26.8 (5.29)
ALSAQ-40 Total Score [Mean (Standard Deviation); unit: score on a scale] — ALSAQ-40 = Amyotrophic Lateral Sclerosis Assessment Questionnaire; summary scores range from 0 (best health status) to 100 (worst health status); ALSAQ-40 total score is calculated as the sum of the summary scores from the 5 domains; lower score corresponds to better health-related quality of life. Population: Full Analysis Set was used.
  score on a scale
    number analyzed (Participants) | 323 | 159 | 482
    (all) | 29.1 (15.56) | 31.6 (16.80) | 29.9 (16.00)
Average Maximum Handgrip Strength [Mean (Standard Deviation); unit: pounds] — Population: Full Analysis Set was used.
  pounds
    number analyzed (Participants) | 323 | 159 | 482
    (all) | 40.22 (26.122) | 38.28 (26.439) | 39.58 (26.216)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Reldesemtiv Versus Placebo on Functional Outcomes in Amyotrophic Lateral Sclerosis (ALS)
Description: Change from baseline to Week 24 in Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) total score using MMRM without multiple imputation; rating scale 0 to 48; higher scores indicate better functional status
Time Frame: Baseline to Week 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reldesemtiv Group, Double-Blind Period | Placebo Group, Double-Blind Period
Number analyzed (Participants) | 323 | 159
score on a scale | -5.57 (5.307) | -4.76 (4.420)

2. Secondary Outcome: Effect of Reldesemtiv Versus Placebo on Combined Functional and Survival Outcomes in Amyotrophic Lateral Sclerosis (ALS)
Description: Composite Assessment of Function and Survival (CAFS) compares ranked outcomes based on change from baseline in ALS Functional Rating Scale-Revised (ALSFRS-R) score (0-48; higher scores indicate better function), time in months to dependence on assisted ventilation (DOAV) and time in months to death. Deceased participants are ranked by time-to-death; earliest deaths ranked the lowest. DOAV survivors are ranked more favorably than those who have died but lower than those alive and not DOAV. Non-DOAV survivors are ranked based on change in ALSFRS-R (largest decline in ALSFRS-R ranked lower than less decline or improvement in ALSFRS-R). Unitless ranked scores range from 1-482 (Full Analysis Set) with larger rank scores associated with a better outcome. Ranks were analyzed using stratified Wilcoxon test comparing the ranked scores between reldesemtiv and placebo, adjusting for baseline riluzole and edaravone use. The win probability and the ratio (reldesemtiv vs placebo) are presented.
Time Frame: Baseline to Week 24
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: unitless
Arm/Group | Reldesemtiv Group, Double-Blind Period | Placebo Group, Double-Blind Period
Number analyzed (Participants) | 323 | 159
unitless | 232.5 [211.0 to 257.0] | 264.0 [209.0 to 291.0]

3. Secondary Outcome: Effect of Reldesemtiv Versus Placebo on Ventilatory Function
Description: Change from baseline in percent predicted forced vital capacity (FVC) using an in-clinic spirometer; a negative number for change from baseline indicates respiratory function decline relative to baseline
Time Frame: Baseline to Week 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Reldesemtiv Group, Double-Blind Period | Placebo Group, Double-Blind Period
Number analyzed (Participants) | 323 | 159
percent predicted | -10.562 (12.8178) | -9.677 (13.1073)

4. Secondary Outcome: Effect of Reldesemtiv Versus Placebo on Quality of Life
Description: Change from baseline in ALSAQ-40 total score. ALSAQ-40 = Amyotrophic Lateral Sclerosis Assessment Questionnaire; summary scores range from 0 (best health status) to 100 (worst health status); ALSAQ-40 total score is calculated as the sum of the summary scores from the 5 domains; lower score corresponds to better health-related quality of life.
Time Frame: Baseline to Week 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reldesemtiv Group, Double-Blind Period | Placebo Group, Double-Blind Period
Number analyzed (Participants) | 323 | 159
score on a scale | 11.426 (12.2102) | 9.766 (11.3662)

5. Secondary Outcome: Effect of Reldesemtiv Versus Placebo on Handgrip Strength
Description: Change from baseline in maximum handgrip strength (average of both hands) measured bilaterally by an electronic hand dynamometer
Time Frame: Baseline to Week 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Reldesemtiv Group, Double-Blind Period | Placebo Group, Double-Blind Period
Number analyzed (Participants) | 323 | 159
pounds | -10.134 (9.6821) | -7.370 (9.7733)

ADVERSE EVENTS:
Time Frame: up to 48 weeks
Arm/Group | Reldesemtiv Group, Double-Blind Period | Placebo Group, Double-Blind Period | Delayed Start Group, Active Drug Period | Early Start Group, Active Drug Period
All-Cause Mortality (participants affected / at risk) | 9/325 | 6/161 | 5/96 | 8/180
Serious Adverse Events (participants affected / at risk) | 41/325 | 25/161 | 14/96 | 33/180
Other Adverse Events (participants affected / at risk) | 258/325 | 125/161 | 65/96 | 122/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reldesemtiv Group, Double-Blind Period (N=325) | Placebo Group, Double-Blind Period (N=161) | Delayed Start Group, Active Drug Period (N=96) | Early Start Group, Active Drug Period (N=180)
pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3) | 4 (4) | 7 (7)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
dysphagia (Gastrointestinal disorders) | 6 (6) | 5 (5) | 2 (2) | 8 (8)
intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
systemic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
vascular device infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
vital capacity decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
refeeding syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
amyotropic lateral sclerosis (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
motor neurone disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
cerebellar stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
assisted suicide (Psychiatric disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
device malfunction (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
mechanical ventilation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
euthanasia (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
medical device change (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reldesemtiv Group, Double-Blind Period (N=325) | Placebo Group, Double-Blind Period (N=161) | Delayed Start Group, Active Drug Period (N=96) | Early Start Group, Active Drug Period (N=180)
COVID-19 (Infections and infestations) | 30 (30) | 13 (13) | 8 (8) | 12 (12)
urinary tract infection (Infections and infestations) | 20 (20) | 9 (9) | 6 (6) | 13 (13)
nasopharyngitis (Infections and infestations) | 17 (17) | 6 (6) | 3 (3) | 2 (2)
fall (Injury, poisoning and procedural complications) | 58 (58) | 23 (23) | 12 (12) | 27 (27)
constipation (Gastrointestinal disorders) | 26 (26) | 12 (12) | 3 (3) | 10 (10)
nausea (Gastrointestinal disorders) | 24 (24) | 6 (6) | 2 (2) | 6 (6)
diarrhoea (Gastrointestinal disorders) | 22 (22) | 14 (14) | 4 (4) | 13 (13)
headache (Nervous system disorders) | 25 (25) | 13 (13) | 7 (7) | 6 (6)
dizziness (Nervous system disorders) | 14 (14) | 8 (8) | 1 (1) | 2 (2)
alanine aminotransferase increased (Investigations) | 21 (21) | 3 (3) | 5 (5) | 3 (3)
aspartate aminotransferase increased (Investigations) | 18 (18) | 1 (1) | 5 (5) | 2 (2)
fatigue (General disorders) | 18 (18) | 10 (10) | 2 (2) | 3 (3)
arthralgia (Musculoskeletal and connective tissue disorders) | 19 (19) | 10 (10) | 3 (3) | 9 (9)
contusion (Injury, poisoning and procedural complications) | 12 (12) | 6 (6) | 2 (2) | 11 (11)
dysphagia (Gastrointestinal disorders) | 7 (7) | 6 (6) | 2 (2) | 9 (9)

LIMITATIONS AND CAVEATS:
The Data Monitoring Committee reviewed unblinded data at the second planned interim analysis and recommended discontinuation of the clinical trial due to futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT04944784/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT04944784/SAP_001.pdf